CLINICAL TRIAL: NCT06679751
Title: Massachusetts HIV and Justice Involved Populations Research Network
Brief Title: Infectious Disease (ID) Testing OUtreach in Carceral Hubs
Acronym: ID-TOUCH
Status: Recruiting | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); South Bay House of Corrections (Unknown); Nashua Street Jail (Unknown)
Responsible Party: Sponsor
Other Study IDs: H-45426; 1R61DA060588-01 (NIH)
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections; Opioid Use Disorder
Keywords: Carceral system; HIV testing; Pre-exposure prophylaxis (PrEP); Justice Community Opioid Innovation Network (JCOIN); End HIV Epidemic (EHE); HIV Services
MeSH Terms: conditions — HIV Infections; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ID-TOUCH Program: Participants will receive the ID-TOUCH intervention while incarcerated and meet with the study team three times for data collection: once before release, once one week after release, and once three months after release. Information collected will include: utilization of HIV services while in jail and while in the community and an exploration of self-reported high-risk behavior, perceived stigma and discrimination, and medical mistrust.
  Interventions: Behavioral: ID-TOUCH

INTERVENTIONS:
Behavioral: ID-TOUCH — ID TOUCH is a multi-pronged intervention to increase HIV testing and PrEP linkage that includes jail-based HIV care process improvements with post-incarceration outreach and linkage to community services.

SUMMARY:
This pilot feasibility study represents part 3 of a larger R61 study, where the investigators will follow a cohort about their experiences with human immunodeficiency virus (HIV) testing.

This project aims to assess the effectiveness of an intervention at two jail sites in the Boston area: South Bay House of Corrections and Nashua Street Jail implemented in January of 2025 that is aimed at improving HIV testing practices and HIV treatment in those carceral facilities. This implementation was developed independently of the investigators' study activities. The jails worked to develop changes in their electronic health record to offer HIV testing at various points in their intake and physical exam process. HIV care was not well-integrated with the jails' existing intake and healthcare administration systems and medications for opioid use disorder (MOUD) program. The investigators will evaluate the intervention the jails developed to address these issues. The outcomes of interest are more implementation than effectiveness outcomes.

The primary goal of this study is to identify existing barriers in the carceral healthcare setting that prevent the improvement of HIV testing and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Incarcerated at South Bay House of Corrections or Nashua Street Jail
* Participant Report that they will be leaving jail within 1 month.
* Participant must be comfortable speaking in the English Language
* Has Opioid Use Disorder (OUD) indicated by participation in Medications for Opioid Use Disorder (MOUD) program and/or self-report

Exclusion Criteria:

* Cognitive ability that prevents obtained consent or completion of study activities (defined through Research Assistant (RA) determination)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are currently incarcerated in either South Bay Correctional Facility or Nashua Street Jail. To be considered eligible they must have opioid use disorder (OUD), be older than 18 years of age, and by self-report say that they will be released from the jail within about one month of the day of study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants that use HIV services while incarcerated | on average 4-6 weeks
  This will be assessed from a review of information abstracted from study questionnaires and interviews with study staff and recorded as a binary 'Yes or No'. If there is any mention of HIV services of any type such as testing, obtaining information. or counseling related to HIV while incarcerated, the participant will be categorized as using HIV services/Yes.
Number of participants that use of PrEP if HIV negative | 1 week, 3 months post incarceration
  This will be assessed from a review of information abstracted from study questionnaires and interviews with study staff and recorded as a binary 'Yes or No'. For participants who are HIV negative, if there is any mention of PrEP being used the participant will be categorized as using PrEP/Yes.
Number of participants that have HIV testing in the community if unknown status during incarceration | 1 week, 3 months post incarceration
  This will be assessed from a review of information abstracted from study questionnaires and interviews with study staff and recorded as a binary 'Yes or No'. Participants with unknown HIV status during incarceration who are tested for HIV in the community, will be categorized as Yes.

SECONDARY OUTCOMES:
Number of participants that demonstrate HIV knowledge | 1 week, 3 months post incarceration
  This will be assessed from a review of information abstracted from study questionnaires and interviews with study staff and recorded as a binary 'Yes or No'. Participants who demonstrate HIV knowledge will be categorized as Yes.
Number of participants that have Risk Behaviors for HIV | 1 week, 3 months post incarceration
  This will be assessed from a review of information abstracted from study questionnaires and interviews with study staff and recorded as a binary 'Yes or No'. Participants who have rsk behaviors for HIV will be categorized as Yes.
Number of participants that have substance use | 1 week, 3 months post incarceration
  This will be assessed from a review of information abstracted from study questionnaires and interviews with study staff and recorded as a binary 'Yes or No'. Participants who report they use substances [eg smoking cigarettes, drinking alcohol, or using any illicit drugs] will be categorized as Yes.
Number of participants with Sexually Transmitted infections (STIs) | 1 month, 3 months post incarceration
  This will be assessed from a review of information abstracted from study questionnaires and interviews with study staff and recorded as a binary 'Yes or No'. Participants who report that they were tested and told they have any STI other than HIV [eg syphilis, gonorrhea, hepatitis C virus (HCV)] will be categorized as Yes.
Number of participants with PrEP Awareness | 1 week, 3 months post incarceration
  This will be assessed from a review of information abstracted from study questionnaires and interviews with study staff and recorded as a binary 'Yes or No'. Participants who demonstrate awareness about PrEP will be categorized as Yes.
Number of participants with acute healthcare utilization | 1 week, 3 months post incarceration
  This will be assessed from a review of information abstracted from study questionnaires and interviews with study staff and recorded as a binary 'Yes or No'. Participants who report they were either hospitalized or received care in an emergency room will be categorized as Yes.

CONTACTS AND LOCATIONS:
Overall Officials: Alysse Wurcel, MD MS, Principal Investigator — Boston Medical Center
Locations (1):
- South Bay House of Corrections, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No